CLINICAL TRIAL: NCT04023838
Title: Randomized Comparison of Radiation Exposure in Coronary Angiography Between Right Conventional and Left Distal Radial Artery Approach: The DOSE Trial
Brief Title: Randomized Comparison of Radiation Exposure in Coronary Angiography Between Right Conventional and Left Distal Radial Artery Approach
Acronym: DOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Myung Ho Jeong, Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DOSE
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Radiation Exposure; Vascular Access Complication; Radial Artery Injury
Keywords: Radiation; Snuffbox approach; Radial approach; Vascular access

STUDY DESIGN:
Intervention Model Description: Patients will be randomized either conventional right radial approach or left distal radial approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right conventional radial approach (Placebo Comparator): After local anesthesia on right wrist area with lidocaine hydrochloride using a 26 gauge needle, the puncture is performed using a 20 gauge needle with the through-and-through puncture technique or a 21 gauge open needle with anterior wall puncture technique. After the successful puncture, 0.025-inch straight wire or 0.018-inch hair wire are inserted, followed by insertion of the 5Fr. radial sheath (Prelude® Radial; Merit medical, UT, USA or Radifocus® Introducer II or Glidesheath Slender®; Terumo Corporation, Tokyo, Japan).
  Interventions: Procedure: artery puncture and coronary angiography
- Left distal radial approach (Active Comparator): After local anesthesia on left anatomical snuffbox area with lidocaine hydrochloride using a 26 gauge needle, the puncture is performed using a 20 gauge needle with the through-and-through puncture technique or a 21 gauge open needle with anterior wall puncture technique. After the successful puncture, 0.025-inch straight wire or 0.018-inch hair wire are inserted, followed by insertion of the 5Fr. radial sheath (Prelude® Radial; Merit medical, UT, USA or Radifocus® Introducer II or Glidesheath Slender®; Terumo Corporation, Tokyo, Japan).
  Interventions: Procedure: artery puncture and coronary angiography

INTERVENTIONS:
Procedure: artery puncture and coronary angiography — We will perform coronary angiography through a Judkins 5 French diagnostic catheter and will take a basic view. At the end of the examination, the radial sheath is removed and the right conventional radial approach is performed for about 4 hours and the left snuffbox approach for about 2 hours using the compressive bandage method. The hemostatic device will use ez ClotRadial® (SOYEON medical Co., Ltd., Wonju, Korea).

SUMMARY:
Randomized comparison of radiation exposure in coronary angiography between right conventional and left distal radial artery approach

DETAILED DESCRIPTION:
The left snuffbox approach is expected to be easier to perform because of less severe tortuosity of the clavicle artery. However, clinical validation of the snuffbox approach was not completed compared with the conventional radial approach. Especially, there is no clinical data on the comparison of the radiation dose in both approaches. To date, there have been some studies on the radiation dose between the left and right radial artery and femoral artery puncture site, but no studies have been conducted on the left snuffbox approach.

The purpose of this study was to compare the radiation doses of the two interventional radiologists by randomly assigning coronary angiography to the left snuffbox approach and right conventional radial approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are a palpable right radial artery and left distal radial artery
* The decision to participate voluntarily in this study and the written consent of the patient

Exclusion Criteria:

* Patients who are not palpable right radial artery and left distal radial artery
* Patients who have arteriovenous fistula
* Patients presenting with acute myocardial infarction
* Patients who need to perform coronary angiography via femoral approach, such as shock state
* Patients who have atrioventricular block on the electrocardiogram
* Patients who have a plan to perform Ergonovine provocation test
* Patients who need percutaneous coronary intervention
* Patients who are not appropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Radiation dose of the operator (µSv) | Through procedure completion, up to 6 hours
  Radiation dose (µSv) of the operator's head, hand, and body will be compared between right conventional radial artery approach and left snuffbox approach group.

SECONDARY OUTCOMES:
Fluoroscopy time for coronary angiography (second) | Through procedure completion, up to 6 hours
  Fluoroscopy time (second) will be compared between two groups during coronary angiography.
Dose-area product (mGy*cm2) | Through procedure completion, up to 6 hours
  Dose-area product (DAP) (mGy*cm2) will be compared between two groups during coronary angiography.
Success rate of radial puncture (%) | Through procedure completion, up to 6 hours
  Successful introduction of sheath (%)
Cannulation time (second) | Through procedure completion, up to 6 hours
  Time from local anesthesia to sheath cannulation (second)
Hemostasis duration (minute) | During hospitalization, up to 1 month
  Hemostasis (minute) is obtained by compressive bandage with ez ClotRadial® (SOYEON medical Co., Ltd., Wonju, Korea)
Puncture site complication after hemostasis | During hospitalization, up to 1 month
  Evaluation of puncture-site bleeding complication using EASY criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, Study Director — Department of Cardiology, Chonnam National University Hospital

IPD SHARING:
Plan to Share IPD: No